CLINICAL TRIAL: NCT00452322
Title: Long-Term Intervention Phase 2 Study of Safety Aspects of Testosterone Undecanoate i.m. in Hypogonadal Men
Brief Title: Safety of Testosterone Undecanoate i.m. in Hypogonadal Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRM 96/17; EK 78a/97Nie1
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2007-03-27 (Estimated); Status verified 2007-03

CONDITIONS: Hypogonadism
Keywords: Testosterone; Hypogonadism; Safety
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Testosterone Substitution by Testosterone Undecanoate i.m.

SUMMARY:
Treatment of male hypogonadism by testosterone substitution has be monitored in terms of safety. This study relates to safety of a new long-acting preparation.

DETAILED DESCRIPTION:
A reliable form of androgen substitution therapy regarding kinetics, tolerance and restoration of androgenicity is paramount in hypogonadal men. Intramuscular injection of the long-acting ester testosterone undecanoate (TU) offers a new modality.

The objective is to assess safety of TU regarding metabolic and pharmacogenetic confounders in hypogonadal men treated with this new formulation.

This is a longitudinal prospective one-arm open intervention and observation trial. A minimum of 5 individual assessments is a prerequisite. Investigated modulators of safety parameters entering regression models are: nadir and/or delta total testosterone concentrations, body mass index (BMI), and age.

The setting Andrological outpatient department.

ELIGIBILITY:
Inclusion Criteria:

* Men presenting hypogonadism-related symptoms and desiring substitution therapy. Such symptoms are fatigue, loss of libido, depressiveness, change in body composition/weight, decreased physical performance, decrease in aggressive behaviour, disability to cope, decreased work performance, lack of androgenization. At least one of these symptoms has to be accompanied by low total testosterone levels (< 12 nmol / L).
* All patients have to give written informed consent for the use of their data for scientific evaluation as approved by the Ethics Committee of the Medical Faculty, University of Muenster, Germany and the State Medical Board.

Exclusion Criteria:

* Prostate Cancer
* Breast Cancer
* Desired Paternity

Ages: 17 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 1997-04; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Prostate (size, PSA-level)
Erythropoeisis (Hemoglobin, Hematocrit)
Lipoproteins (HDL, LDL, Triglycerides)
Blood pressure
Pulse

SECONDARY OUTCOMES:
Possible changes of body mass index

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard Nieschlag, MD, PhD, Study Director — University Clinics Muenster, Germany
Locations (1):
- Institute of Reproductive Medicine of the University Clinics, Münster, Germany

REFERENCES:
- [Derived] Zitzmann M, Nieschlag E. Androgen receptor gene CAG repeat length and body mass index modulate the safety of long-term intramuscular testosterone undecanoate therapy in hypogonadal men. J Clin Endocrinol Metab. 2007 Oct;92(10):3844-53. doi: 10.1210/jc.2007-0620. Epub 2007 Jul 17. PMID 17635942